CLINICAL TRIAL: NCT04362397
Title: Foco: Evaluating a Training to Increase Attention and Awareness in the Daily Activities of Healthcare Professionals
Brief Title: FoCo: Evaluating a Training to Increase Attention and Awareness of Healthcare Professionals
Acronym: FoCo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: HIAE_FoCo
Record Dates: First submitted 2019-12-19; First posted 2020-04-24 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2019-12

CONDITIONS: Attention; Self-compassion

STUDY DESIGN:
Intervention Model Description: Group A will receive training in the FoCo program and group B will be a waiting list group. After a period of one month, group B will receive training in FoCo and group A will be instructed to continue on their own to apply FoCo in their daily lives.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator responsible for the statistical analysis will be blind to the groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (first group to receive the intervention) (Experimental): This arm will receive the attention, care, and self-care training first.
  Interventions: Behavioral: FoCo; Behavioral: No intervention
- B (second group to receive the intervention) (Experimental): This arm will not receive intervention in the first month and will receive it after this period.
  Interventions: Behavioral: FoCo; Behavioral: No intervention

INTERVENTIONS:
Behavioral: FoCo — This is an attention, care and self-care training.
Behavioral: No intervention — This is a waiting list

SUMMARY:
Introduction: A significant increase in the risk of injury and illness at work has been associated with fatigue, stress, haste, distraction, emergency situations, excessive noise, complex procedures and anger among other factors.

Most of these factors are related to the lack of attention to work in progress, which can be improved by training attention and awareness during daily activities, as it would encourage a resumption of focus on the task at hand and the possible risks associated with it. . The primary objective of this project is to evaluate the effects of training to increase attention and awareness for daily activities - FoCo - outlined for healthcare professionals in their work schedule. Method: Health professionals from 18 to 60 years of age, of both sexes, will participate in the study, working in 3 units, one in the care of patients in a Emergency Care Unit (UPA), in an Elderly Residential and in a Center. Intensive Care (ICU). In the UPA will be included 25 professionals in group A and 25 in group B; In the Residential of Elderly, 40 professionals will be included in group A and 40 professionals in group B; In the ICU will be included 30 professionals in group A and 30 in group B. They will be randomized in both groups. Group A will receive training in the FoCo program and group B will be a waiting group. After a period of one month, group B will receive training in FoCo and group A will be instructed to continue on their own to apply FoCo in their daily lives (Fig.1). Participants will be evaluated before, after one month and after two months. Expected Outcomes: After training, an increase in mindful, attention and awareness scale, self-compassion scale, positive affect, speed of digit and symbol test is expected. It is also expected to reduce negative affects, perceived stress and an increased perception of possible incidents.

ELIGIBILITY:
Inclusion Criteria:

* be available to participate in the training and to perform the evaluations before and after it.

Exclusion Criteria:

- being away or on vacation during the research project, being in psychiatric treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
change in stress | 1 month
  The authors will evaluate attention using the MAAS (Mindful Attention Awareness Scale).
change in attention | 1 month
  The authors will apply the Perceived Stress Scale

SECONDARY OUTCOMES:
change in self-compassion | 1 month
  The authorswill apply the self-compassion scale
change in sleep | 1 month
  The authors will apply the Pittsburgh inventory
change in Mental health symptoms | 1 month
  The authors will apply the SRQ-20 (self-report questionnaire)
change in positive and negative affect | 1 month
  The authors will apply PANAS

CONTACTS AND LOCATIONS:
Overall Officials: Elisa H Kozasa, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No